CLINICAL TRIAL: NCT06146751
Title: A Novel Ferumoxytol-enhanced Cardiac Magnetic Resonance Imaging for the Detection of Intracardiac Thrombus in Patients With Ventricular Aneurysm and After Percutaneous Ventricular Reconstruction
Brief Title: A Novel Ferumoxytol-enhanced Cardiac Magnetic Resonance Imaging for the Detection of Intracardiac Thrombus
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Chunjian Li, Dr., MD, PhD, Deputy Director, Department of Cardiology; Director, Coronary Care Unit, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: 024
Record Dates: First submitted 2023-11-18; First posted 2023-11-27 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Heart Aneurysm
Keywords: ferumoxytol; ultrasmall superparamagnetic iron oxide particles; contrast-enhanced magnetic resonance; thrombosis; ventricular aneurysm
MeSH Terms: conditions — Heart Aneurysm; Thrombosis | interventions — Magnetic Iron Oxide Nanoparticles; Ferrosoferric Oxide

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with ventricular aneurysm and after percutaneous ventricular reconstruction: Patients with ventricular aneurysm and after percutaneous ventricular reconstruction undergo a novel ferumoxytol-enhanced cardiac magnetic resonance imaging and transthoracic echocardiography.
  Interventions: Drug: Superparamagnetic Iron Oxide Nanoparticles

INTERVENTIONS:
Drug: Superparamagnetic Iron Oxide Nanoparticles — Patients will receive a novel ferumoxytol-enhanced cardiac magnetic resonance imaging.
  Other Names: ferumoxytol

SUMMARY:
The incidence of thrombosis in ventricular aneurysm was reported to be 35%-40%, which may lead to systemic thromboembolism. Patients with ventricular aneurysm without detectable thrombus are not routinely treated with anticoagulation. Therefore, the accuracy of intracardiac thrombus detection has an important impact on clinical management decisions. Currently, transthoracic echocardiography is the most commonly used method to detect intracardiac thrombus, but its sensitivity and positive predictive value are low. Cardiac magnetic resonance has a higher diagnostic accuracy for intracardiac thrombus, and its sensitivity and positive predictive value are higher than those of transthoracic echocardiography and CT. However, the gadolinium-based contrast agents commonly used for enhanced magnetic resonance imaging have some problems such as nephrogenic systemic fibrosis, gadolinium deposition in the brain, and short imaging time. Ferumoxytol, a superparamagnetic iron oxide nanoparticle, can be used for off-label enhanced magnetic resonance imaging. Its long intravascular half-life makes it suitable for enhanced magnetic resonance imaging with complex scanning procedures and long repetitive scans. Ferumoxytol is cleared from the blood pool by macrophages of the reticuloendothelial system, mainly in the spleen and lymph nodes. Therefore, ferumoxytol has a favourable safety even in adults and children with end-stage renal failure. The aim of this study is to evaluate the effectiveness of a novel ferumoxytol-enhanced cardiac magnetic resonance in detecting intracardiac thrombus in patients with ventricular aneurysm and after percutaneous ventricular reconstruction.

DETAILED DESCRIPTION:
Ferumoxytol is a member of ultrasmall superparamagnetic iron oxide particles with an average diameter of 30 nm, originally developed as an intravascular contrast agent for MRI. Ferumoxytol was approved by the FDA in 2009 for the intravenous treatment of iron deficiency anaemia in adults with chronic kidney disease, and has also been used off-label as a non-gadolinium contrast agent for whole-body magnetic resonance imaging. Its iron oxide core is coated with dextran, which reduces immunogenicity and delays phagocytosis and the release of elemental iron from the core. As a result, ferumoxytol has a long intravascular half-life of approximately 15 hours and is slowly taken up by the macrophages of the reticuloendothelial system. Because of its long half-life, ferumoxytol is suitable for enhanced magnetic resonance imaging with complex scanning procedures and long repetitive scans. Ferumoxytol has been proved to be safe even in adults and children with end-stage renal failure. As feraheme is not available in the Chinese market, we experimentally synthesised a new formulation of ferumoxytol, which is identical to ferumoxytol in terms of physicochemical structure, pharmacokinetics and toxicological effects, at the request of Chia Tai Tianqing Pharmaceutical Group Co, Ltd (Nanjing, China) in 2014. This study is a single-centre, prospective, observational, non-randomised study. The study will enrol patients with ventricular aneurysm and after percutaneous ventricular reconstruction. The aim of this study is to evaluate the effectiveness of ferumoxytol-enhanced cardiac magnetic resonance imaging in detecting intracardiac thrombus in patients with ventricular aneurysm and left ventricular thrombus in the dynamic chamber and static chamber in patients 180±30 days after percutaneous ventricular reconstruction by comparing the detection rate of intracardiac thrombus with ferumoxytol-enhanced cardiac magnetic resonance imaging and transthoracic echocardiography, and to provide a clinical basis for the development and application of the new generation of magnetic resonance contrast agents in China. The echocardiography and magnetic resonance imaging experts were blinded to each other's results.

ELIGIBILITY:
Inclusion criteria:

1. Age ≥ 18 years and ≤ 80 years;
2. Patients with left ventricular aneurysm detected by transthoracic echocardiography or 180±30 days after percutaneous ventricular reconstruction;
3. An informed consent form was signed voluntarily by the patients or an authorised family member.

Exclusion criteria:

1. Patients unable to lie down for any reason;
2. Patients who are unable to undergo MRI for psychological (e.g. suffering from claustrophobia syndrome) or physical reasons (e.g. non-antimagnetic metal retention in the body, hearing impairment, involuntary body movements, etc.);
3. Patients with a known history of iron allergy or hypersensitivity;
4. Patients taking other oral or intravenous iron products;
5. Patients with haemosiderin deposition or haemochromatosis;
6. Pregnant or lactating women;
7. Any other patient that the investigator deems inappropriate for enrolment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 patients with ventricular aneurysm and 10 to 20 patients after percutaneous ventricular reconstruction at the First Affiliated Hospital of Nanjing Medical University
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
detection rate of intracardiac thrombus | Nov. 1st, 2023 to Mar. 31st, 2025
  Detection rate of intracardiac thrombus by ferumoxytol-enhanced magnetic resonance and transthoracic echocardiography
detection rate of thrombus in dynamic chamber and static chamber | Nov. 1st, 2023 to Mar. 31st, 2025
  Detection rate of thrombus in dynamic chamber and static chamber by ferumoxytol-enhanced magnetic resonance and transthoracic echocardiography in patients after percutaneous ventricular reconstruction

CONTACTS AND LOCATIONS:
Overall Officials: Chunjian Li, MD, PhD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Delewi R, Zijlstra F, Piek JJ. Left ventricular thrombus formation after acute myocardial infarction. Heart. 2012 Dec;98(23):1743-9. doi: 10.1136/heartjnl-2012-301962. No abstract available. PMID 23151669
- [Background] El Ouazzani J, Jandou I. Aneurysm and pseudoaneurysm of the left ventricle. Ann Med Surg (Lond). 2022 Feb 24;75:103405. doi: 10.1016/j.amsu.2022.103405. eCollection 2022 Mar. PMID 35386778
- [Background] Ibanez B, James S, Agewall S, Antunes MJ, Bucciarelli-Ducci C, Bueno H, Caforio ALP, Crea F, Goudevenos JA, Halvorsen S, Hindricks G, Kastrati A, Lenzen MJ, Prescott E, Roffi M, Valgimigli M, Varenhorst C, Vranckx P, Widimsky P; ESC Scientific Document Group. 2017 ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation: The Task Force for the management of acute myocardial infarction in patients presenting with ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2018 Jan 7;39(2):119-177. doi: 10.1093/eurheartj/ehx393. No abstract available. PMID 28886621
- [Background] O'Gara PT, Kushner FG, Ascheim DD, Casey DE Jr, Chung MK, de Lemos JA, Ettinger SM, Fang JC, Fesmire FM, Franklin BA, Granger CB, Krumholz HM, Linderbaum JA, Morrow DA, Newby LK, Ornato JP, Ou N, Radford MJ, Tamis-Holland JE, Tommaso CL, Tracy CM, Woo YJ, Zhao DX, Anderson JL, Jacobs AK, Halperin JL, Albert NM, Brindis RG, Creager MA, DeMets D, Guyton RA, Hochman JS, Kovacs RJ, Kushner FG, Ohman EM, Stevenson WG, Yancy CW; American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. 2013 ACCF/AHA guideline for the management of ST-elevation myocardial infarction: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. Circulation. 2013 Jan 29;127(4):e362-425. doi: 10.1161/CIR.0b013e3182742cf6. Epub 2012 Dec 17. No abstract available. PMID 23247304
- [Background] Whalen H, Dako F, Patel P, Sahbaz J, Hong-Zohlman S, White CS, Jeudy J. Role of Imaging for Suspected Cardiac Thrombus. Curr Treat Options Cardiovasc Med. 2019 Dec 9;21(12):81. doi: 10.1007/s11936-019-0792-6. PMID 31820132
- [Background] Allard L, Bernhard B, Windecker S, Valgimigli M, Grani C. Left ventricular thrombus in ischaemic heart disease: diagnosis, treatment, and gaps of knowledge. Eur Heart J Qual Care Clin Outcomes. 2022 Aug 17;8(5):496-509. doi: 10.1093/ehjqcco/qcab097. PMID 34928322
- [Background] Srichai MB, Junor C, Rodriguez LL, Stillman AE, Grimm RA, Lieber ML, Weaver JA, Smedira NG, White RD. Clinical, imaging, and pathological characteristics of left ventricular thrombus: a comparison of contrast-enhanced magnetic resonance imaging, transthoracic echocardiography, and transesophageal echocardiography with surgical or pathological validation. Am Heart J. 2006 Jul;152(1):75-84. doi: 10.1016/j.ahj.2005.08.021. PMID 16824834
- [Background] Wertman R, Altun E, Martin DR, Mitchell DG, Leyendecker JR, O'Malley RB, Parsons DJ, Fuller ER 3rd, Semelka RC. Risk of nephrogenic systemic fibrosis: evaluation of gadolinium chelate contrast agents at four American universities. Radiology. 2008 Sep;248(3):799-806. doi: 10.1148/radiol.2483072093. Epub 2008 Jul 15. PMID 18632533
- [Background] Sadowski EA, Bennett LK, Chan MR, Wentland AL, Garrett AL, Garrett RW, Djamali A. Nephrogenic systemic fibrosis: risk factors and incidence estimation. Radiology. 2007 Apr;243(1):148-57. doi: 10.1148/radiol.2431062144. Epub 2007 Jan 31. PMID 17267695
- [Background] Kribben A, Witzke O, Hillen U, Barkhausen J, Daul AE, Erbel R. Nephrogenic systemic fibrosis: pathogenesis, diagnosis, and therapy. J Am Coll Cardiol. 2009 May 5;53(18):1621-8. doi: 10.1016/j.jacc.2008.12.061. PMID 19406336
- [Background] Stojanov D, Aracki-Trenkic A, Benedeto-Stojanov D. Gadolinium deposition within the dentate nucleus and globus pallidus after repeated administrations of gadolinium-based contrast agents-current status. Neuroradiology. 2016 May;58(5):433-41. doi: 10.1007/s00234-016-1658-1. Epub 2016 Feb 12. PMID 26873830
- [Background] Roberts DR, Holden KR. Progressive increase of T1 signal intensity in the dentate nucleus and globus pallidus on unenhanced T1-weighted MR images in the pediatric brain exposed to multiple doses of gadolinium contrast. Brain Dev. 2016 Mar;38(3):331-6. doi: 10.1016/j.braindev.2015.08.009. Epub 2015 Sep 4. PMID 26345358
- [Background] Hu HH, Pokorney A, Towbin RB, Miller JH. Increased signal intensities in the dentate nucleus and globus pallidus on unenhanced T1-weighted images: evidence in children undergoing multiple gadolinium MRI exams. Pediatr Radiol. 2016 Oct;46(11):1590-8. doi: 10.1007/s00247-016-3646-3. Epub 2016 Jun 9. PMID 27282825
- [Background] Finn JP, Nguyen KL, Hu P. Ferumoxytol vs. Gadolinium agents for contrast-enhanced MRI: Thoughts on evolving indications, risks, and benefits. J Magn Reson Imaging. 2017 Sep;46(3):919-923. doi: 10.1002/jmri.25580. Epub 2017 Feb 3. No abstract available. PMID 28160356
- [Background] Finn JP, Nguyen KL, Han F, Zhou Z, Salusky I, Ayad I, Hu P. Cardiovascular MRI with ferumoxytol. Clin Radiol. 2016 Aug;71(8):796-806. doi: 10.1016/j.crad.2016.03.020. Epub 2016 May 21. PMID 27221526
- [Background] Neuwelt EA, Hamilton BE, Varallyay CG, Rooney WR, Edelman RD, Jacobs PM, Watnick SG. Ultrasmall superparamagnetic iron oxides (USPIOs): a future alternative magnetic resonance (MR) contrast agent for patients at risk for nephrogenic systemic fibrosis (NSF)? Kidney Int. 2009 Mar;75(5):465-74. doi: 10.1038/ki.2008.496. Epub 2008 Oct 8. PMID 18843256
- [Background] Nayak AB, Luhar A, Hanudel M, Gales B, Hall TR, Finn JP, Salusky IB, Zaritsky J. High-resolution, whole-body vascular imaging with ferumoxytol as an alternative to gadolinium agents in a pediatric chronic kidney disease cohort. Pediatr Nephrol. 2015 Mar;30(3):515-21. doi: 10.1007/s00467-014-2953-x. Epub 2014 Sep 12. PMID 25212105
- [Background] Muehe AM, Feng D, von Eyben R, Luna-Fineman S, Link MP, Muthig T, Huddleston AE, Neuwelt EA, Daldrup-Link HE. Safety Report of Ferumoxytol for Magnetic Resonance Imaging in Children and Young Adults. Invest Radiol. 2016 Apr;51(4):221-227. doi: 10.1097/RLI.0000000000000230. PMID 26656202
- [Background] Wang YX, Idee JM. A comprehensive literatures update of clinical researches of superparamagnetic resonance iron oxide nanoparticles for magnetic resonance imaging. Quant Imaging Med Surg. 2017 Feb;7(1):88-122. doi: 10.21037/qims.2017.02.09. PMID 28275562
- [Background] Li W, Salanitri J, Tutton S, Dunkle EE, Schneider JR, Caprini JA, Pierchala LN, Jacobs PM, Edelman RR. Lower extremity deep venous thrombosis: evaluation with ferumoxytol-enhanced MR imaging and dual-contrast mechanism--preliminary experience. Radiology. 2007 Mar;242(3):873-81. doi: 10.1148/radiol.2423052101. PMID 17325072
- [Background] Dong Z, Si G, Zhu X, Li C, Hua R, Teng J, Zhang W, Xu L, Qian W, Liu B, Wang J, Wang T, Tang Y, Zhao Y, Gong X, Tao Z, Xu Z, Li Y, Chen B, Kong X, Xu Y, Gu N, Li C. Diagnostic Performance and Safety of a Novel Ferumoxytol-Enhanced Coronary Magnetic Resonance Angiography. Circ Cardiovasc Imaging. 2023 Jul;16(7):580-590. doi: 10.1161/CIRCIMAGING.123.015404. Epub 2023 Jul 18. PMID 37463240
- [Background] Toth GB, Varallyay CG, Horvath A, Bashir MR, Choyke PL, Daldrup-Link HE, Dosa E, Finn JP, Gahramanov S, Harisinghani M, Macdougall I, Neuwelt A, Vasanawala SS, Ambady P, Barajas R, Cetas JS, Ciporen J, DeLoughery TJ, Doolittle ND, Fu R, Grinstead J, Guimaraes AR, Hamilton BE, Li X, McConnell HL, Muldoon LL, Nesbit G, Netto JP, Petterson D, Rooney WD, Schwartz D, Szidonya L, Neuwelt EA. Current and potential imaging applications of ferumoxytol for magnetic resonance imaging. Kidney Int. 2017 Jul;92(1):47-66. doi: 10.1016/j.kint.2016.12.037. Epub 2017 Apr 20. PMID 28434822
- [Background] Lehrman ED, Plotnik AN, Hope T, Saloner D. Ferumoxytol-enhanced MRI in the peripheral vasculature. Clin Radiol. 2019 Jan;74(1):37-50. doi: 10.1016/j.crad.2018.02.021. Epub 2018 May 3. PMID 29731126